CLINICAL TRIAL: NCT06309888
Title: Magnetic Resonance Imaging of Cognitive Deficits in the Brain of Individuals With Spinal Cord Injury
Acronym: SCI_Cog
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2023-18
Record Dates: First submitted 2024-01-26; First posted 2024-03-13 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; neuroimaging; cognition; executive functions
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- spinal cord injury: Individuals living with a spinal cord injury
- non spinal cord injury: able-bodied individuals

SUMMARY:
In the case of spinal cord injury, rehabilitation is particularly focused on motor skills. Non-motor impairments such as thinking difficulties did not receive a lot of attention to date.

In this research project, the investigators want to find out how thinking difficulties become noticeable in the brain with spinal cord injury.

Participation procedure: Participants who take part will be asked to come to an examination once. The duration of the examination is between 2 and 2.5 hours (including around 55 minutes in the magnetic resonance imaging scanner, including preparation and follow-up).

ELIGIBILITY:
Inclusion criteria (with and without spinal cord injury):

* Male or Female
* Age between 18 and 60
* German native speaker
* Normal or corrected-to-normal visual acuity

Additional inclusion criteria (spinal cord injury only):

* A diagnosis of traumatic spinal cord injury (SCI)
* Time since injury 12 months or longer
* American Spinal Injury Association Impairment Scale (AIS) grade A, B, C and D

Exclusion criteria (with and without spinal cord injury):

* Contraindication for magnetic resonance imaging examinations (e.g., cardiac pacemaker etc.)
* Pregnancy
* Diagnosis of other psychiatric or neurological disorders (including tumor in the central nervous system)
* Alcohol and/or drug abuse
* Confirmed diagnosis of traumatic brain injury
* Insufficient hand function (not able to hold a pen due to the restricted motor abilities)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals with SCI and healthy controls will be recruited for the study considering age-matching.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Brain activity | Baseline
  Brain activity defined as changes in oxygen levels in the blood during the execution of cognitive tasks on cognitive inhibition and verbal fluency (executive functions), and at rest

SECONDARY OUTCOMES:
Behavioral performance | Baseline
  Accuracy on cognitive inhibition task (in percentage)
Behavioral performance | Baseline
  Reaction time (in milliseconds) on cognitive inhibition task
Behavioral performance | Baseline
  Number of errors on cognitive inhibition task
Behavioral performance | Baseline
  Number of correct words on verbal fluency task
Behavioral performance | Baseline
  Number of mistakes on verbal fluency task
Brain morphometry | Baseline
  Volume of brain structures in cubic millimetres
Level of life satisfaction | Baseline
  Satisfaction with Life Scale (validated questionnaire assessing life satisfaction)
Level of anxiety | Baseline
  State-Trait Anxiety Inventory (validated questionnaire assessing anxiety)
Level of pain | Baseline
  Validated questionnaire assessing pain severity
Quality of sleep | Baseline
  Pittsburgh Sleep Quality Index (validated questionnaire assessing sleep quality)
Level of attention and awareness | Baseline
  Mindful Attention and Awareness scale (validated questionnaire assessing level of attention and awareness)
Motor symptom severity | Baseline
  Motor symptoms severity (from level A to E) based on the International Standards for Neurological Classification of spinal cord injury (ISNCSCI)
Demographics | Baseline
  Demographic information such as age, sex and education level, as well as time since injury

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Research, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No
The investigators plan to save anonymised data into public repositories, but given the size of imaging data, they are still undecided.